CLINICAL TRIAL: NCT07168447
Title: Effect of Exchange Transfusions on Cognitive Efficiency in Patients With Sickle Cell Disease
Brief Title: Transfusion Exchanges and Cognition in Sickle Cell Disease
Acronym: DREPA-COG
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D24-P021; IDRCB : 2024-A02851-46 (Other: ANSM)
Record Dates: First submitted 2025-08-18; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Drepanocytosis; Chronic Neurological Deficiency
Keywords: Sickle cell disease; cognitive function; neuropsychological assessment; transfusion exchange; non-interventional study; executive function, SDMT, T-MoCA, fatigue, anxiety, depression
MeSH Terms: conditions — Sickle Cell Trait; Anemia, Sickle Cell; Fatigue; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
DREPA-COG is an observational study evaluating the effect of exchange transfusions on cognitive function in adults with severe sickle cell disease (SS or Sβ0). Information processing speed is assessed at three time points during the transfusion cycle using the Symbol Digit Modalities Test (SDMT) and additional validated neuropsychological measures. This minimal-risk, fully remote study aims to identify processing speed as a reproducible marker for clinical monitoring and future therapeutic trials.

DETAILED DESCRIPTION:
DREPA-COG is a non-interventional, multicenter observational study investigating the effect of exchange transfusions on cognitive performance in adults with severe sickle cell disease (SS or Sβ0). Cognitive complications, including slowed information processing and executive dysfunction, are frequent and disabling in this population. Exchange transfusion, a standard therapy replacing sickled red blood cells with donor cells, may positively influence cognition, but systematic evidence is lacking.

The study evaluates information processing speed as a potential neurological marker across the transfusion cycle. Participants complete three brief neuropsychological assessments remotely by videoconference: before the transfusion, one week after, and prior to the next transfusion. The Symbol Digit Modalities Test (SDMT) is the primary measure, complemented by validated assessments of global cognition, attention, memory, fatigue, mood, and pain.

Primary analysis will use mixed-effects models to assess changes in processing speed over time, adjusting for demographic and clinical covariates. This minimal-risk, fully remote study requires no additional hospital visits and aims to establish processing speed as a reproducible and clinically relevant outcome measure in sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with severe sickle cell disease (SS or Sβ0).
* Enrolled in a regular monthly transfusion exchange program.
* Not institutionalized.
* No known dementia.
* No severe aphasia.
* Affiliated with or beneficiary of a social security system.

Exclusion criteria:

* Insufficient mastery of spoken French.
* Severe comorbidities preventing short-term follow-up.
* Known psychiatric disorders.
* Participation in another clinical study with ongoing exclusion periods.
* Lack of adequate computer equipment (minimum 11-inch screen and internet connection).
* Vulnerable patients under legal protection (guardianship or curatorship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 18 years or older with severe sickle cell disease (SS or Sβ0) who are enrolled in a regular monthly transfusion exchange program. Participants must not be institutionalized, must have no known dementia or severe aphasia, and must be able to communicate in French. They must also be affiliated with a social security system. Excluded are individuals with severe comorbidities that could interfere with short-term follow-up, those with known psychiatric disorders, participants in other ongoing clinical studies with exclusion periods, individuals lacking adequate computer equipment for remote assessments, and vulnerable patients under legal protection such as guardianship or curatorship. This population allows evaluation of cognitive processing speed and other neuropsychological outcomes in a controlled, transfusion-managed cohort of adult sickle cell patients.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2025-12-03 (Estimated); Primary Completion 2027-11-02 (Estimated); Study Completion 2027-11-02 (Estimated)

PRIMARY OUTCOMES:
Information Processing Speed | 48 hours before the transfusion exchange
  Primary outcome measure: Information processing speed, assessed using the oral version of the Symbol Digit Modality Test (SDMT), as a marker of cerebral involvement in adult patients with sickle cell disease.
Information Processing Speed | 7 to 9 days after the transfusion exchange
  Primary outcome measure: Information processing speed, assessed using the oral version of the Symbol Digit Modality Test (SDMT), as a marker of cerebral involvement in adult patients with sickle cell disease.
Information Processing Speed | within 48 hours before the next scheduled transfusion exchange
  Primary outcome measure: Information processing speed, assessed using the oral version of the Symbol Digit Modality Test (SDMT), as a marker of cerebral involvement in adult patients with sickle cell disease.

SECONDARY OUTCOMES:
Global Cognitive Function - Montreal Cognitive Assessment (Telephone version, T-MoCA) | Time Point 1 (Baseline): within 48 hours before the scheduled exchange transfusion. Time Point 2 (Post-transfusion): 7 to 9 days after the exchange transfusion. Time Point 3 (End of cycle): within 48 hours before the next scheduled exchange transfusion
  The T-MoCA is a validated screening tool for global cognition, adapted for telephone administration. Scores range from 0 to 22, with higher scores indicating better cognitive performance.
Fatigue Severity Score (FSS) | Time Point 1 (Baseline): within 48 hours before the scheduled exchange transfusion. Time Point 2 (Post-transfusion): 7 to 9 days after the exchange transfusion. Time Point 3 (End of cycle): within 48 hours before the next scheduled exchange transfusion
  Fatigue will be assessed using the Fatigue Severity Scale (FSS), a validated self-administered questionnaire consisting of 9 items, each rated on a 7-point Likert scale (1 = strongly disagree; 7 = strongly agree).
  The total score is the mean of the 9 items, ranging from 1 (no fatigue) to 7 (severe fatigue).
  Higher scores indicate more severe fatigue and represent a worse outcome.
Anxiety and Depression Symptoms (Hospital Anxiety and Depression Scale, HADS | Time Point 1 (Baseline): within 48 hours before the scheduled exchange transfusion. Time Point 2 (Post-transfusion): 7 to 9 days after the exchange transfusion. Time Point 3 (End of cycle): within 48 hours before the next scheduled exchange transfusion
  The Hospital Anxiety and Depression Scale (HADS) is a validated self-report questionnaire consisting of 14 items, divided into two subscales: Anxiety (HADS-A, 7 items) and Depression (HADS-D, 7 items). Each subscale score ranges from 0 to 21, with higher scores indicating more severe symptoms.
Pain Intensity (Numeric Rating Scale, NRS) | Time Point 1 (Baseline): within 48 hours before the scheduled exchange transfusion. Time Point 2 (Post-transfusion): 7 to 9 days after the exchange transfusion. Time Point 3 (End of cycle): within 48 hours before the next scheduled exchange transfusion
  Pain intensity will be assessed using the Numeric Rating Scale (NRS), a validated self-report tool where participants rate their pain on a scale from 0 to 10.
  0 = no pain
  10 = worst imaginable pain Higher scores indicate greater pain intensity.
Change in Information Processing Speed Measured by the Symbol Digit Modalities Test (SDMT) | Within 48 hours before exchange transfusion 7-9 days after exchange transfusion Within 48 hours before the next scheduled exchange transfusion
  Information processing speed will be assessed using the Symbol Digit Modalities Test (SDMT), a standardized neuropsychological test that evaluates attention, visual scanning, and motor speed. The test provides a raw score, which reflects the number of correct pairings completed within a 90-second period.
  Higher scores indicate better information processing speed.
  This measure aims to evaluate changes in SDMT scores across the transfusion cycle and identify individual variability in performance.
Working Memory - WAIS-IV Digit Span Subtest | Time Point 1 (Baseline): within 48 hours before the scheduled exchange transfusion. Time Point 2 (Post-transfusion): 7 to 9 days after the exchange transfusion. Time Point 3 (End of cycle): within 48 hours before the next scheduled exchange transfusion
  The Digit Span subtest from the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV), assesses working memory capacity. Scores range from 0 to 16, with higher scores reflecting better performance.

CONTACTS AND LOCATIONS:
Overall Officials: HUGO BISMUTH, DOCTOR, Principal Investigator — Hôpital Sainte-Anne; David CLAVET, PROFESSOR, Study Chair — Hôpital Sainte-Anne
Locations (6):
- France (6):
  - Assistance Publique - Hôpitaux de Paris Hôpital Avicenne, Bobigny, Île-de-France Region
  - Hôpital Henri Mondor, Créteil, Île-de-France Region
  - Hôpital Kremlin-Bicêtre, Le Kremlin-Bicêtre, Île-de-France Region
  - GHU Paris Psychiatrie et Neurosciences - Hôpital Sainte-Anne, Paris, Île-de-France Region
  - Assistance Publique - Hôpitaux de Paris Hôpital Necker, Paris, Île-de-France Region
  - Centre Hospitalier Saint-Denis, Saint-Denis, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-07-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT07168447/Prot_000.pdf